CLINICAL TRIAL: NCT04997837
Title: A Multicenter, Randomized, Controlled Phase III Study of Chemotherapy With or Without PD-1 Inhibitors and Chemoradiotherapy as Adjuvant Regimen for D2/R0 Resected pN3 Gastric (G) or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Study of Adjuvant Chemotherapy With or Without PD-1 Inhibitors and Chemoradiotherapy in Resected pN3 Gastric (G) or GEJ Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2021-63-2366
Record Dates: First submitted 2021-07-21; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immune Checkpoint Inhibitors; Oxaliplatin; Capecitabine; Fluorouracil; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor and chemoradiotherapy (Experimental): PD-1 inhibitor+CapeOX/SOX/FOLFOX for 6 weeks, followed by chemoradiotherapy; 6 weeks of PD-1 inhibitor and CapeOX/SOX/FOLFOX for 6 weeks after chemoradiotherapy, followed by PD-1 inhibitor, till 12 months after chemoradiotherapy.
  PD-1 inhibitor Nivolumab/Toripalimab 240mg solution intravenously once daily, Q2W. OR Nivolumab/Toripalimab 360mg solution intravenously once daily, Q3W; OR Pembrolizumab/Tilelizumab/Sintilimab/Carrelizumab, 200mg solution intravenously once daily, Q3W.
  Chemotherapy: CapeOx or SOX or FOLFOX therapy determined by investigator.
  Chemoradiotherapy Radiotherapy: 1.8 Gy/fx, 45-50.5Gy Chemotherapy: Capecitabine 625mg/m2 bid orally with radiotherapy; OR Tegafur-gimeracil-oteracil potassium combination drug 40-60mg bid orally with radiotherapy.
  Interventions: Drug: PD-1 inhibitor; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Tegafur-gimeracil-oteracil potassium; Drug: 5-FU; Radiation: Radiotherapy; Drug: Chemotherapy
- Chemotherapy (Active Comparator): Chemotherapy: CapeOx or SOX or FOLFOX therapy determined by investigator.
  CapeOX:
  Oxaliplatin 130 mg/m2 (body surface area) solution intravenously once-daily, followed by 20 days off.
  Capecitabine 1000 mg2 (body surface area) bid orally in 14 days, followed by 7 days off.
  SOX:
  Oxaliplatin 130 mg/m2 (body surface area) solution intravenously once-daily, followed by 20 days off.
  Tegafur-gimeracil-oteracil potassium combination drug 40 - 60 mg bid orally in 14 days, followed by 7 days off.
  FOLFOX:
  Oxaliplatin 85 mg/m2 (body surface area) solution intravenously once-daily, followed by 13 days off.
  5-FU 2400-2800mg/m2/d continuous intravenous pumping for 48h, Q2W.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Tegafur-gimeracil-oteracil potassium; Drug: 5-FU

INTERVENTIONS:
Drug: PD-1 inhibitor — Nivolumab/Toripalimab 240mg solution intravenously once daily, Q2W. OR Nivolumab/Toripalimab 360mg solution intravenously once daily, Q3W; OR Pembrolizumab/Tilelizumab/Sintilimab/Carrelizumab, 200mg solution intravenously once daily, Q3W.
  Arms: PD-1 inhibitor and chemoradiotherapy
Drug: Oxaliplatin — CapeOx: 130 mg/m2 (body surface area) solution intravenously once-daily, followed by 20 days off.
  FOLFOX: 85 mg/m2 (body surface area) solution intravenously once-daily, followed by 13 days off.
Drug: Capecitabine — CapeOx: 1000 mg2 (body surface area) bid orally in 14 days, followed by 7 days off.
Drug: Tegafur-gimeracil-oteracil potassium — SOX: 40 - 60 mg bid orally in 14 days, followed by 7 days off
Drug: 5-FU — FOLFOX：2400-2800mg/m2/d continuous intravenous pumping for 48h, Q2W
Radiation: Radiotherapy — 1.8 Gy/Fx, 45-50.4 Gy
  Arms: PD-1 inhibitor and chemoradiotherapy
Drug: Chemotherapy — Capecitabine 625mg/m2 bid orally with radiotherapy; ORegafur-gimeracil-oteracil potassium combination drug 40-60mg bid orally with radiotherapy
  Arms: PD-1 inhibitor and chemoradiotherapy

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of postoperative adjuvant chemotherapy with PD-1 inhibitors and chemoradiotherapy, in comparison with adjuvant chemotherapy only, in D2/R0 resected pN3 gastric or gastroesophageal junction adenocarcinoma. PD-1+CRT cohort: A total of 216 patients will receive 6 weeks of PD-1 inhibitors and chemotherapy, then receive concurrent chemoradiotherapy, followed by 6 weeks of PD-1 inhibitors and chemotherapy, finally receive maintenance treatment of PD-1 inhibitors until (maximum 1year after radiotherapy). CT cohort: A total of 217 patients will receive 6 months of chemotherapy. The disease-free survival(DFS), overall survival(OS) and adverse effects will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1
* Patients with expected survival time more than 6 months
* Patients after standard D2/R0 resection
* Postoperative histologically confirmed adenocarcinoma of the stomach or GEJ
* Positive lymph nodes more than 7, stage pN3
* Patients without distant metastasis (M0) or M1 with abdominal exfoliated cell detection positive (CY1P0)
* Patients' physical condition and visceral function allows following adjuvant therapy, including chemotherapy, chemoradiotherapy and PD-1 inhibitor therapy.
* Patients' blood routine and biochemical indicators should meet the following standard: Hb≥90g/L, ANC≥1.5*10^9/L, PLT≥100*10^9/L, ALT & AST≤2.5 U/L, TB ≤ 1.5 UNL, serum creatinine<1 UNL.
* Patients who are willing to obey regimens during the study.
* Written informed consent is acquired before random entry, and patients should know that he/she has the right to quit, and following treatment won't be affected.
* Patients are willing to provide samples of blood and tissue.

Exclusion Criteria:

* Patients with gross peritoneal metastasis (CY1P0 excluded) or distant metastasis.
* Patients who has received any anti-tumor therapy before surgery.
* Patients who had received radiotherapy for abdominal organs including stomach, liver, kidney, etc.
* Patients who had active systematic autoimmune diseases which need systematic treatment within 2 years before first medication in the study, substitutive therapy (such as thyroxine, insulin, etc) excluded.
* Patients diagnosed with immunodeficiency, or was receiving systematic glucocorticoid treatment or other immunosuppressive therapy within 7 days before medication, physiological dose of glucocorticoid is allowed (≤10 mg/d prednison or equivalent medication)
* Patients who have known severe allergic reaction (≥level 3) to anti-PD-1 monoclonal antibody, 5-FU, Oxaliplatin or any auxiliary material.
* Patient diagnosed with other malignant tumor in the past 5 years, excluding radical basal cell carcinoma of the skin and/or radical resected carcinoma in situ.
* Patient with severe vital organ failure.
* Pregnant or lactation period
* Patient with known mental illness or drug abuse that may influence compliance.
* Patient with known HIV infection, or active tuberculosis.
* Untreated active hepatitis B
* Patient with active HCV infection
* Uncontrolled complications
* Other situations that might disturb study results and compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
3-year DFS rate | Up to 3 years
  Defined as the time from randomization to the date of first documented progression or death from any cause.

SECONDARY OUTCOMES:
3-year OS rate | Up to 3 years
  Defined as the time from randomization to death from any cause.
3-year local recurrence free survival rate | Up to 3 years
  Defined as the time from randomization to the date of first documented recurrence or death from any cause.
Percentage of participants with treatment-related acute adverse events as assessed by CTCAE v5.0 | Up to 28 days from last dose
Quality of life as assessed by Quality of Life Scale (range 0-60) | Through study completion, up to 10 years
  It evaluates the quality of life from 12 aspects, including appetite, mental status, sleep quality, fatigue, etc. The higher scores mean a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yang W, Zhou M, Li G, Zhou C, Wang L, Xia F, Zhang H, Shen L, Wang Y, Wan J, Wang Y, Zhao G, Zhang Z. Adjuvant chemoradiotherapy plus PD-1 inhibitor for pN3 gastric cancer: a randomized, multicenter, Phase III trial. Future Oncol. 2024 Dec;20(40):3389-3396. doi: 10.1080/14796694.2024.2421156. Epub 2024 Nov 15. PMID 39545610